CLINICAL TRIAL: NCT00979875
Title: Phase 1, Randomized, Double-Blind, Pharmacokinetic and Glucodynamic, 6-Way Crossover Study of Subcutaneously Administered Insulin Analogs With Recombinant Human Hyaluronidase (rHuPH20) Compared to Insulin Analogs Alone in Healthy Volunteers
Brief Title: A Pharmacokinetic and Glucodynamic Study of Subcutaneously Administered Insulin Analogs With rHuPH20 Compared to Insulin Analogs Alone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: HALO-117-104
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: insulin; recombinant human hyaluronidase; Healthy volunteers
MeSH Terms: conditions — Insulin Resistance | interventions — Insulin Lispro; insulin glulisine; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lispro+PH20, Lispro, Glulis+PH20, Glulis, Aspart+PH20, Aspart (Experimental): All participants were randomized to 1 of 6 treatment sequences (ABC, ACB, BAC, BCA, CAB, or CBA), each of which was comprised of the same 3 interventions (A, B, and C). Each intervention was separated by a 3- to 14-day washout.
  Intervention A: Participants received a single, subcutaneous (SC) injection of 95 units per milliliter (U/mL) Lispro + 5 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20 (PH20) and a single, SC injection of 95 U/mL Lispro alone 3 to 14 days apart.
  Intervention B: Participants received a single, SC injection of 95 U/mL Glulisine (Glulis) + 5 µg/mL PH20 and a single, SC injection of 95 U/mL Glulis alone 3 to 14 days apart.
  Intervention C: Participants received a single, SC injection of 95 U/mL Aspart + 5 µg/mL PH20 and a single, SC injection of 95 U/mL Aspart alone 3 to 14 days apart.
  Interventions: Drug: Recombinant human hyaluronidase PH20 (rHuPH20); Drug: Insulin lispro; Drug: Insulin glulisine; Drug: Insulin aspart

INTERVENTIONS:
Drug: Recombinant human hyaluronidase PH20 (rHuPH20)
  Other Names: HYLENEX; PH20
Drug: Insulin lispro
  Other Names: Humalog; Lispro
Drug: Insulin glulisine
  Other Names: Apidra; Glulisine
Drug: Insulin aspart
  Other Names: NovoLog; Aspart

SUMMARY:
This is a single-center, Phase 1, randomized, double-blind, 6-way crossover study to determine insulin pharmacokinetics, insulin glucodynamics, safety, and tolerability of subcutaneously administered dose(s) of insulin lispro + recombinant human hyaluronidase PH20 (rHuPH20), insulin lispro alone, insulin glulisine + rHuPH20, insulin glulisine alone, insulin aspart + rHuPH20, and insulin aspart alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants between the ages of 18 and 55 years, inclusive (healthy is defined as no clinically relevant abnormalities).
* Body mass index (BMI) between 18-27 kilograms per meter squared (kg/m^2), inclusive.
* Total body weight >65 kilograms (kg) (143 pounds [lb]) for men and >46 kg (101 lb) for women.
* Decision making capacity and willingness to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures including adequate venous access.
* Vital signs (blood pressure [BP], pulse rate, body temperature) within normal range or, if out of range, assessed by the Principal Investigator as not clinically significant.
* Fasting blood glucose level <100 milligrams per deciliter (mg/dL) at screening.
* A negative serum pregnancy test (if female of childbearing potential).
* Female participants of childbearing potential must agree to practice effective birth control or abstinence currently and agree to continue to do so for the duration of their time on study.
* Signed, written institutional review board (IRB)-approved informed consent.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, oncologic, or neurologic (to include history of seizures) disease; hypoglycemic episodes; intercurrent illness (such as influenza); or allergic disease (including severe drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing). Clinical significance to be determined by the Principal Investigator.
* As judged by the investigator, clinically significant findings in routine laboratory data. (Anemia with hematocrit less than 33% at screening is specifically exclusionary.)
* Known history of diabetes mellitus (type 1 or type 2) or gestational diabetes.
* Known allergy to hyaluronidase or any other ingredient in the study drug.
* Positive human immunodeficiency virus (HIV) 1, hepatitis B, or hepatitis C antibody test.
* History or evidence of alcohol or drug abuse.
* History or evidence of use of any tobacco- or nicotine-containing product within 6 months prior to screening and a screening qualitative urine nicotine test.
* Use of drugs that may interfere with the interpretation of study results or are known to cause clinically relevant interference with insulin action or glucose utilization.
* Blood donation or high volume phlebotomy, for example, >100 milliliters (mL), within 56 days before dosing.
* Participation in a study of any investigational drug or device 30 days before enrollment in this study.
* The participant is unfit for the study in the opinion of the investigator.
* Women who are pregnant or breast-feeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Hompesch, M.D., Principal Investigator — Profil Institute for Clinical Research, Inc.
Locations (1):
- Profil Institute for Clinical Research, Inc., Chula Vista, California, United States

REFERENCES:
- [Derived] Morrow L, Muchmore DB, Hompesch M, Ludington EA, Vaughn DE. Comparative pharmacokinetics and insulin action for three rapid-acting insulin analogs injected subcutaneously with and without hyaluronidase. Diabetes Care. 2013 Feb;36(2):273-5. doi: 10.2337/dc12-0808. Epub 2012 Oct 5. PMID 23043164

RESULTS

PARTICIPANT FLOW:
Groups:
- Lispro+PH20, Lispro, Glulis, Glulis+PH20, Aspart, Aspart+PH20: Participants received a single, subcutaneous (SC) injection of 95 units per milliliter (U/mL) Lispro + 5 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20 (PH20). Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Lispro alone.
  After a 3- to 14-day washout, participants received a single, SC injection of 95 U/mL Glulisine (Glulis) alone. Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Glulis + 5 µg/mL PH20.
  After a 3- to 14-day washout, participants received a single, SC injection of 95 U/mL Aspart alone. Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Aspart + 5 µg/mL PH20.
- Glulis+PH20, Glulis, Lispro+PH20, Lispro, Aspart+PH20, Aspart: Participants received a single, subcutaneous (SC) injection of 95 units per milliliter (U/mL) Glulisine (Glulis) + 5 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20 (PH20). Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Glulis alone.
  After a 3- to 14-day washout, participants received a single, SC injection of 95 U/mL Lispro + 5 µg/mL PH20. Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Lispro alone.
  After a 3- to 14-day washout, participants received a single, SC injection of 95 U/mL Aspart + 5 µg/mL PH20. Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Aspart alone.
- Lispro, Lispro+PH20, Aspart, Aspart+PH20, Glulis, Glulis+PH20: Participants received a single, subcutaneous (SC) injection of 95 units per milliliter (U/mL) Lispro alone. Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Lispro + 5 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20 (PH20).
  After a 3- to 14-day washout, participants received a single, SC injection of 95 U/mL Aspart alone. Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Aspart + 5 µg/mL PH20.
  After a 3- to 14-day washout, participants received a single, SC injection of 95 U/mL Glulisine (Glulis) alone. Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Glulis + 5 µg/mL PH20.
- Glulis, Glulis+PH20, Aspart+PH20, Aspart, Lispro+PH20, Lispro: Participants received a single, subcutaneous (SC) injection of 95 units per milliliter (U/mL) Glulisine (Glulis) alone. Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Glulis + 5 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20 (PH20).
  After a 3- to 14-day washout, participants received a single, SC injection of 95 U/mL Aspart + 5 µg/mL PH20. Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Aspart alone.
  After a 3- to 14-day washout, participants received a single, subcutaneous (SC) injection of 95 U/mL Lispro + 5 µg/mL PH20. Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Lispro alone.
- Aspart+PH20, Aspart, Glulis+PH20, Glulis, Lispro, Lispro+PH20: Participants received a single, subcutaneous (SC) injection of 95 units per milliliter (U/mL) Aspart + 5 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20 (PH20). Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Aspart alone.
  After a 3- to 14-day washout, participants received a single, SC injection of 95 U/mL Glulisine (Glulis) + 5 µg/mL PH20. Then, 3 to 14 days later, participants received and a single, SC injection of 95 U/mL Glulisine alone.
  After a 3- to 14-day washout, participants received a single, SC injection of 95 U/mL Lispro alone. Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Lispro + 5 µg/mL PH20.
- Aspart, Aspart+PH20, Lispro, Lispro+PH20, Glulis+PH20, Glulis: Participants received a single, subcutaneous (SC) injection of 95 units per milliliter (U/mL) Aspart alone. Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Aspart + 5 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20 (PH20).
  After a 3- to 14-day washout, participants received a single, SC injection of 95 U/mL Lispro alone. Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Lispro + 5 µg/mL PH20.
  After a 3- to 14-day washout, participants received a single, SC injection of 95 U/mL Glulisine (Glulis) + 5 µg/mL PH20. Then, 3 to 14 days later, participants received a single, SC injection of 95 U/mL Glulis alone.
Period: Intervention 1
Arm/Group | Lispro+PH20, Lispro, Glulis, Glulis+PH20, Aspart, Aspart+PH20 | Glulis+PH20, Glulis, Lispro+PH20, Lispro, Aspart+PH20, Aspart | Lispro, Lispro+PH20, Aspart, Aspart+PH20, Glulis, Glulis+PH20 | Glulis, Glulis+PH20, Aspart+PH20, Aspart, Lispro+PH20, Lispro | Aspart+PH20, Aspart, Glulis+PH20, Glulis, Lispro, Lispro+PH20 | Aspart, Aspart+PH20, Lispro, Lispro+PH20, Glulis+PH20, Glulis
Started | 2 | 2 | 3 | 2 | 3 | 2
Received at Least 1 Dose of Study Drug | 2 | 2 | 3 | 2 | 3 | 2
Completed | 2 | 2 | 3 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 1 (3 to 14 Days)
Arm/Group | Lispro+PH20, Lispro, Glulis, Glulis+PH20, Aspart, Aspart+PH20 | Glulis+PH20, Glulis, Lispro+PH20, Lispro, Aspart+PH20, Aspart | Lispro, Lispro+PH20, Aspart, Aspart+PH20, Glulis, Glulis+PH20 | Glulis, Glulis+PH20, Aspart+PH20, Aspart, Lispro+PH20, Lispro | Aspart+PH20, Aspart, Glulis+PH20, Glulis, Lispro, Lispro+PH20 | Aspart, Aspart+PH20, Lispro, Lispro+PH20, Glulis+PH20, Glulis
Started | 2 | 2 | 3 | 2 | 3 | 2
Completed | 2 | 2 | 3 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 2
Arm/Group | Lispro+PH20, Lispro, Glulis, Glulis+PH20, Aspart, Aspart+PH20 | Glulis+PH20, Glulis, Lispro+PH20, Lispro, Aspart+PH20, Aspart | Lispro, Lispro+PH20, Aspart, Aspart+PH20, Glulis, Glulis+PH20 | Glulis, Glulis+PH20, Aspart+PH20, Aspart, Lispro+PH20, Lispro | Aspart+PH20, Aspart, Glulis+PH20, Glulis, Lispro, Lispro+PH20 | Aspart, Aspart+PH20, Lispro, Lispro+PH20, Glulis+PH20, Glulis
Started | 2 | 2 | 3 | 2 | 3 | 2
Completed | 2 | 2 | 3 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 2 (3 to 14 Days)
Arm/Group | Lispro+PH20, Lispro, Glulis, Glulis+PH20, Aspart, Aspart+PH20 | Glulis+PH20, Glulis, Lispro+PH20, Lispro, Aspart+PH20, Aspart | Lispro, Lispro+PH20, Aspart, Aspart+PH20, Glulis, Glulis+PH20 | Glulis, Glulis+PH20, Aspart+PH20, Aspart, Lispro+PH20, Lispro | Aspart+PH20, Aspart, Glulis+PH20, Glulis, Lispro, Lispro+PH20 | Aspart, Aspart+PH20, Lispro, Lispro+PH20, Glulis+PH20, Glulis
Started | 2 | 2 | 3 | 2 | 3 | 2
Completed | 2 | 2 | 3 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 3
Arm/Group | Lispro+PH20, Lispro, Glulis, Glulis+PH20, Aspart, Aspart+PH20 | Glulis+PH20, Glulis, Lispro+PH20, Lispro, Aspart+PH20, Aspart | Lispro, Lispro+PH20, Aspart, Aspart+PH20, Glulis, Glulis+PH20 | Glulis, Glulis+PH20, Aspart+PH20, Aspart, Lispro+PH20, Lispro | Aspart+PH20, Aspart, Glulis+PH20, Glulis, Lispro, Lispro+PH20 | Aspart, Aspart+PH20, Lispro, Lispro+PH20, Glulis+PH20, Glulis
Started | 2 | 2 | 3 | 2 | 3 | 2
Completed | 2 | 2 | 3 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Overall Study: All participants were randomized to 1 of 6 treatment sequences (ABC, ACB, BAC, BCA, CAB, or CBA), each of which was comprised of the same 3 interventions (A, B, and C). Each intervention was separated by a 3- to 14-day washout.
  Intervention A: Participants received a single, subcutaneous (SC) injection of 95 units per milliliter (U/mL) Lispro + 5 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20 (PH20) and a single, SC injection of 95 U/mL Lispro alone 3 to 14 days apart.
  Intervention B: Participants received a single, SC injection of 95 U/mL Glulisine (Glulis) + 5 µg/mL PH20 and a single, SC injection of 95 U/mL Glulis alone 3 to 14 days apart.
  Intervention C: Participants received a single, SC injection of 95 U/mL Aspart + 5 µg/mL PH20 and a single, SC injection of 95 U/mL Aspart alone 3 to 14 days apart.
Arm/Group | Overall Study
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve for Serum Insulin From Time 0 to 60 Minutes (AUC0-60)
Description: Area under the concentration (AUC)-time curve was derived as the area under the serum insulin concentration profile from 0 to 60 minutes. Blood samples were taken 30, 20, and 10 minutes (mins) prior to each injection; every 3 mins (from 0 to 15 mins); and at 20, 25, 30, 45, and 60 mins after each injection.
Time Frame: Predose up to 60 minutes postdose
Population: Participants who received at least one dose of Lispro alone, Lispro + recombinant human hyaluronidase PH20 (rHuPH20), Glulisine alone, Glulisine + rHuPH20, Aspart alone, or Aspart + rHuPH20 with evaluable AUC0-60 data.
Measure: Mean (Standard Deviation); unit: minutes*nanomolars (min*nM)
Groups:
- Glulisine Alone: Participants received a single, subcutaneous injection of 95 units per milliliter (U/mL) Glulisine alone.
- Glulisine + rHuPH20: Participants received a single, subcutaneous injection of 95 units per milliliter (U/mL) Glulisine + 5 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20 (rHuPH20).
- Lispro Alone: Participants received a single, subcutaneous injection of 95 units per milliliter (U/mL) Lispro alone.
- Lispro + rHuPH20: Participants received a single, subcutaneous injection of 95 units per milliliter (U/mL) Lispro + 5 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20 (rHuPH20).
- Aspart Alone: Participants received a single, subcutaneous injection of 95 units per milliliter (U/mL) Aspart alone.
- Aspart + rHuPH20: Participants received a single, subcutaneous injection of 95 units per milliliter (U/mL) Aspart + 5 micrograms per milliliter (µg/mL) recombinant human hyaluronidase PH20 (rHuPH20).
Arm/Group | Glulisine Alone | Glulisine + rHuPH20 | Lispro Alone | Lispro + rHuPH20 | Aspart Alone | Aspart + rHuPH20
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
minutes*nanomolars (min*nM) | 11667.14 (4085.00) | 23807.14 (6657.73) | 10687.14 (5532.49) | 27850.00 (9684.94) | 8065.00 (3138.37) | 20778.57 (6383.05)
Statistical Analysis 1: Comparison: Glulisine Alone vs Glulisine + rHuPH20; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Statistical testing was considered exploratory, with no adjustment for inflation of Type 1 error due to multiplicity of testing; Analysis performed using mixed model with fixed effect for treatment. A compound symmetry covariance matrix among repeated measurements was assumed; Geometric Least Squares Mean Ratio = 2.08, 90% CI 2-sided [1.70 to 2.55]
Statistical Analysis 2: Comparison: Lispro Alone vs Lispro + rHuPH20; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares Means Ratio = 5.26, 90% CI 2-sided [3.88 to 7.12]
Statistical Analysis 3: Comparison: Aspart Alone vs Aspart + rHuPH20; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares Means Ratio = 4.14, 90% CI 2-sided [3.05 to 5.60]

2. Secondary Outcome: Time to Maximum Serum Insulin Concentration (Tmax)
Description: Tmax was determined as the timepoint where the maximum of all valid concentration measurements for each measurement series was observed. Samples were taken 30, 20, 10 minutes (mins) prior to each injection; every 3 mins (from 0 to 15 mins); every 5 mins (from 15 to 30 mins); every 15 mins (from 30 to 90 mins); every 30 mins (from 90 to 240 mins); and every 60 mins (from 240 to 480 mins) after each injection.
Time Frame: Predose up to 480 minutes postdose
Population: Participants who received at least one dose of Lispro alone, Lispro + recombinant human hyaluronidase PH20 (rHuPH20), Glulisine alone, Glulisine + rHuPH20, Aspart alone, or Aspart + rHuPH20 with evaluable tmax data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Glulisine Alone | Glulisine + rHuPH20 | Lispro Alone | Lispro + rHuPH20 | Aspart Alone | Aspart + rHuPH20
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
minutes | 80.36 (25.38) | 41.43 (12.47) | 67.50 (32.09) | 41.07 (17.56) | 85.71 (35.99) | 43.57 (12.92)
Statistical Analysis 1: Comparison: Glulisine Alone vs Glulisine + rHuPH20; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = -38.93, 90% CI 2-sided [-53.31 to -24.55]
Statistical Analysis 2: Comparison: Lispro Alone vs Lispro + rHuPH20; Test type: Superiority or Other; p = 0.0032, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = -26.43, 90% CI 2-sided [-40.81 to -12.05]
Statistical Analysis 3: Comparison: Aspart Alone vs Aspart + rHuPH20; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = -42.14, 90% CI 2-sided [-56.53 to -27.76]

3. Secondary Outcome: Time to Early and Late 50% Maximum Serum Insulin Concentration (t[50%Max])
Description: Blood samples were taken 30, 20, 10 minutes (mins) prior to each injection; every 3 mins (from 0 to 15 mins); every 5 mins (from 15 to 30 mins); every 15 mins (from 30 to 90 mins); every 30 mins (from 90 to 240 mins); and every 60 mins (from 240 to 480 mins) after each injection.
Time Frame: Predose up to 480 minutes postdose
Population: Participants who received at least one dose of Lispro alone, Lispro + recombinant human hyaluronidase PH20 (rHuPH20), Glulisine alone, Glulisine + rHuPH20, Aspart alone, or Aspart + rHuPH20 with evaluable t(50%max) data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Glulisine Alone | Glulisine + rHuPH20 | Lispro Alone | Lispro + rHuPH20 | Aspart Alone | Aspart + rHuPH20
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
minutes
  early t(50%max) | 21.06 (9.60) | 10.16 (4.90) | 30.69 (12.58) | 18.96 (5.27) | 31.93 (8.15) | 17.98 (5.22)
  late t(50%max) | 195.43 (48.63) | 118.92 (33.57) | 176.79 (30.00) | 89.59 (21.38) | 193.50 (45.94) | 102.82 (24.74)

4. Secondary Outcome: Time to Maximum Glucose Infusion Rate (tGIR[Max])
Description: as for outcome 3
Time Frame: Predose up to 480 minutes postdose
Population: Participants who received at least one dose of Lispro alone, Lispro + recombinant human hyaluronidase PH20 (rHuPH20), Glulisine alone, Glulisine + rHuPH20, Aspart alone, or Aspart + rHuPH20 with evaluable tGIR(max) data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Glulisine Alone | Glulisine + rHuPH20 | Lispro Alone | Lispro + rHuPH20 | Aspart Alone | Aspart + rHuPH20
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
minutes | 141.93 (71.18) | 113.36 (69.85) | 160.14 (71.36) | 103.57 (58.83) | 158.79 (52.34) | 96.93 (56.65)

5. Secondary Outcome: Percentage of Total Area Under the Concentration-time Curve for Serum Insulin Attained by Time t (AUC0-t)
Description: Percentage of total area under the concentration (AUC)-time curve at 15, 30, 60, 120 minutes after injection was measured. Blood samples were taken 30, 20, 10 minutes (mins) prior to each injection; every 3 mins (from 0 to 15 mins); every 5 mins (from 15 to 30 mins); every 15 mins (from 30 to 90 mins); and at 90 and 120 mins after each injection.
Time Frame: Predose up to 120 minutes postdose
Population: Participants who received at least one dose of Lispro alone, Lispro + recombinant human hyaluronidase PH20 (rHuPH20) , Glulisine alone, Glulisine + rHuPH20, Aspart alone, or Aspart + rHuPH20 with evaluable AUC0-t data.
Measure: Mean (Standard Deviation); unit: percentage of total AUC
Arm/Group | Glulisine Alone | Glulisine + rHuPH20 | Lispro Alone | Lispro + rHuPH20 | Aspart Alone | Aspart + rHuPH20
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
percentage of total AUC
  AUC0-15 | 2.02 (1.10) | 5.29 (2.06) | 0.68 (0.65) | 2.38 (1.24) | 0.56 (0.30) | 2.92 (2.28)
  AUC0-30 | 7.09 (3.40) | 15.82 (5.56) | 3.88 (2.71) | 13.81 (5.37) | 3.54 (1.90) | 13.66 (7.05)
  AUC0-60 | 20.68 (8.07) | 39.45 (10.64) | 18.72 (7.74) | 42.88 (8.89) | 16.85 (6.54) | 41.51 (12.06)
  AUC0-120 | 50.35 (12.69) | 71.70 (11.07) | 50.14 (12.10) | 77.00 (7.54) | 47.97 (12.32) | 77.37 (8.80)

6. Secondary Outcome: Time to Percentage of Total Insulin Exposure
Description: Time to 10% and 50% of total insulin exposure was measured. Samples were taken 30, 20, 10 minutes (mins) prior to each injection; every 3 mins (from 0 to 15 mins); every 5 mins (from 15 to 30 mins); every 15 mins (from 30 to 90 mins); every 30 mins (from 90 to 240 mins); and every 60 mins (from 240 to 480 mins) after each injection.
Time Frame: Predose up to 480 minutes postdose
Population: Participants who received at least one dose of Lispro alone, Lispro + rHuPH20, Glulisine alone, Glulisine + recombinant human hyaluronidase PH20 (rHuPH20), Aspart alone, or Aspart + rHuPH20 with evaluable total insulin exposure data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Glulisine Alone | Glulisine + rHuPH20 | Lispro Alone | Lispro + rHuPH20 | Aspart Alone | Aspart + rHuPH20
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
minutes
  Time to 10% of total insulin exposure | 39.59 (9.95) | 23.39 (6.38) | 46.56 (11.89) | 26.35 (5.60) | 48.42 (9.96) | 26.99 (6.57)
  Time to 50% of total insulin exposure | 123.65 (27.48) | 78.64 (18.82) | 123.39 (27.87) | 70.97 (12.61) | 130.86 (30.04) | 72.53 (14.86)

ADVERSE EVENTS:
Arm/Group | Glulisine Alone | Glulisine + rHuPH20 | Lispro Alone | Lispro + rHuPH20 | Aspart Alone | Aspart + rHuPH20
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 2/14 | 2/14 | 3/14 | 2/14 | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glulisine Alone (N=14) | Glulisine + rHuPH20 (N=14) | Lispro Alone (N=14) | Lispro + rHuPH20 (N=14) | Aspart Alone (N=14) | Aspart + rHuPH20 (N=14)
Infusion site anaesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The Organ System includes "administration site conditions."
Infusion site pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The Organ System includes "administration site conditions."
Infusion site abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days